CLINICAL TRIAL: NCT01456949
Title: Sustained Treatment of Paroxysmal Atrial Fibrillation Post-Approval Study (STOP AF PAS)
Acronym: STOP AF PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOP AF PAS
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Atrial Fibrillation (PAF)
Keywords: Atrial fibrillation (AF); Paroxysmal atrial fibrillation (PAF); Arrythmias; Cardiac Arrythmias; Cardiac ablation; Cryoablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): Cryoablation
  Interventions: Device: Medtronic Arctic Front® Cardiac CryoAblation System

INTERVENTIONS:
Device: Medtronic Arctic Front® Cardiac CryoAblation System — Cardiac cryoablation to isolate the pulmonary veins using the Arctic Front® CryoAblation System, with point ablation using the Freezor® Max as needed.
  Other Names: Medtronic CryoCath CryoConsole; Arctic Front® Cardiac CryoAblation Catheter; Arctic Front Advance™ Cardiac CryoAblation Catheter; Freezor® MAX Cardiac CryoAblation Catheter

SUMMARY:
The Post-Approval Study (PAS) is a prospective multi-center, non-randomized, single arm, controlled,unblinded clinical study designed to provide long-term safety and effectiveness of the Arctic Front® Cardiac CryoAblation System.

DETAILED DESCRIPTION:
Safety and effectiveness will be evaluated against pre-specified performance criteria as determined by the sponsor and FDA. The criteria set in this study have been previously used to demonstrate safety and effectiveness in cryoablation and radio-frequency ablation for the treatment of paroxysmal atrial fibrillation.

The analyses of the primary effectiveness objective will take place once all the subjects with a study cryoablation procedure attempt have reached 36 months of follow-up post-cryoablation procedure. The analysis of the primary safety objective will take place once all the subjects with a study cryoablation procedure attempt have reached 12 months of follow-up post-cryoablation procedure. The analyses for the secondary objectives will take place once all subjects with a study cryoablation attempt have reached 36 months of follow-up post-cryoablation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Documented PAF:

   * Diagnosis of paroxysmal atrial fibrillation (PAF), AND
   * 2 or more episodes of AF during the 3 months preceding the consent Date, AND
   * At least 1 episode of AF documented with a tracing within 12 months preceding the consent date.
2. Age 18 years or older
3. Failure for the treatment of AF (effectiveness or intolerance) of at least one membrane active AAD for rhythm control.

Exclusion Criteria:

1. Any previous left atrial (LA) ablation (except permissible retreatment subjects)
2. Any previous LA surgery
3. Current intracardiac thrombus (can be treated after thrombus is resolved)
4. Presence of any pulmonary vein stents
5. Presence of any pre-existing pulmonary vein stenosis
6. Pre-existing hemidiaphragmatic paralysis
7. Anteroposterior LA diameter > 5.5 cm by TTE
8. Presence of any cardiac valve prosthesis
9. Clinically significant mitral valve regurgitation or stenosis
10. Myocardial infarction, PCI / PTCA or coronary artery stenting which occurred during the 3 month interval preceding the Consent Date
11. Unstable angina
12. Any cardiac surgery which occurred during the 3 month interval preceding the Consent Date
13. Any significant congenital heart defect corrected or not (including atrial septal defects or pulmonary vein abnormalities but not including minor PFO)
14. NYHA class III or IV congestive heart failure
15. Left ventricular ejection fraction (LVEF) < 40%
16. 2º (Type II) or 3º atrioventricular block
17. Presence of a permanent pacemaker, biventricular pacemaker, atrial defibrillator or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
18. Brugada syndrome
19. Long QT syndrome
20. Arrhythmogenic right ventricular dysplasia
21. Sarcoidosis
22. Hypertrophic cardiomyopathy
23. Known cryoglobulinemia
24. Uncontrolled hyperthyroidism
25. Any cerebral ischemic event (strokes or TIAs) which occurred during the 6 month interval preceding the Consent Date.
26. Any woman known to be pregnant
27. Life expectancy less than one (1) year
28. Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of this study not pre-approved by Medtronic
29. Unwilling or unable to comply fully with study procedures and followup

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2012-06-26 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley P. Knight, MD, FACC, FHRS, Principal Investigator — Northwestern Memorial Hospital
Locations (39):
- United States (32):
  - Alaska Heart Institute, Anchorage, Alaska
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Good Samaritan Hospital, San Jose, California
  - Colorado Heart and Vascular, Denver, Colorado
  - Daytona Heart Group, Daytona Beach, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Memorial Advanced Cardiovascular Institute, South Bend, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Metropolitan Cardiology Consultants PA, Coon Rapids, Minnesota
  - St. Mary's Hospital - Mayo Clinic, Rochester, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Bryan LGH, Lincoln, Nebraska
  - Asheville Cardiology Associate PA, Asheville, North Carolina
  - Bethesda North Hospital l TriHealth Hatton Institute, Cincinnati, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Capital Cardiovascular Associates, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Cardiology Associates, Doylestown, Pennsylvania
  - Lancaster Heart & Stroke, Lancaster, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Columbia Heart Clinic, Columbia, South Carolina
  - Stern Cardiovascular, Germantown, Tennessee
  - Saint Thomas Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Saint Luke's Episcopal Hospital - Texas Medical Center, Houston, Texas
  - Baylor Research Institute, Plano, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia
- Canada (7):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials Inc, Victoria, British Columbia
  - Hôpital du Sacre Coeur de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec

REFERENCES:
- [Derived] Knight BP, Novak PG, Sangrigoli R, Champagne J, Dubuc M, Adler SW, Svinarich JT, Essebag V, Hokanson R, Kueffer F, Jain SK, John RM, Mansour M; STOP AF PAS Investigators. Long-Term Outcomes After Ablation for Paroxysmal Atrial Fibrillation Using the Second-Generation Cryoballoon: Final Results From STOP AF Post-Approval Study. JACC Clin Electrophysiol. 2019 Mar;5(3):306-314. doi: 10.1016/j.jacep.2018.11.006. Epub 2018 Dec 26. PMID 30898232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subjects was enrolled on 26 June 2012 and the first study cryoablation occurred on 28 June 2012. The last subject was enrolled on 21 August 2014 and the final study cryoablation occurred on 14 October 2014. As this was a single arm study, all subjects enrolled were planned to have a cryoablation procedure.
Period: Enrollment
Arm/Group | Single Arm
Started | 402
Treated (Enrolled subjects who underwent a study cryoablation procedure whether or not they met I/E criteria.) | 359
Modified Intent to Treat Group (mITT) (Enrolled subjects who met all I/E criteria and underwent a study cryoablation procedure.) | 354
Completed | 365 (6 rollover subjects not included in final analysis. 359 treated; 354 treated & met all I/E criteria.)
Not Completed | 37
Not completed — PI death- incomplete data | 6
Not completed — Death | 1
Not completed — I/E criteria not met prior to procedure | 13
Not completed — Physician Decision | 10
Not completed — Withdrawal by Subject | 7
Period: Study Cryoablation Procedure & Follow-up
Arm/Group | Single Arm
Started | 365
3-month Follow-up Visit Completed | 344 (Of 354 subjects who were treated and met all I/E criteria (mITT group).)
6-month Follow-up Visit Completed | 342 (Of mITT group.)
12-month Follow-up Visit Completed | 325 (Of mITT group.)
24-month Follow-up Visit Completed | 309 (Of mITT group.)
36-month Follow-up Visit Completed | 298 (Of mITT group.)
Completed (Of mITT group.) | 303 (5 subjects completed at least 36 months of follow-up but did not complete a 36 month follow-up visit)
Not Completed | 62
Not completed — Death | 5
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 11
Not completed — Physician Decision | 1
Not completed — Subject Relocation | 10
Not completed — Failure to maintain study compliance | 2
Not completed — Rollover not included in completer total | 6
Not completed — Treated did not meet I/E criteria | 4

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes those subjects who were enrolled and met all inclusion and no exclusions criteria (Intent to Treat population).
Groups:
- Modified Intent to Treat Group (mITT): Enrolled subjects that met all inclusion and no exclusion criteria, and who underwent a study cryoablation procedure.
Arm/Group | Modified Intent to Treat Group (mITT)
Number analyzed (Participants) | 354
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 234
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnic Origin: American Indian or Alaska Native | 1
  Race/Ethnic Origin: Asian | 5
  Race/Ethnic Origin: Black or African American | 1
  Race/Ethnic Origin: Hispanic or Latino | 4
  Race/Ethnic Origin: Native Hawaiian or Pacific Islander | 1
  Race/Ethnic Origin: White or Caucasian | 328
  Race/Ethnic Origin: Other race | 1
  Race/Ethnic Origin: Unknown/Unreported | 13

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness: Percentage of Participants Free of Chronic Treatment Failure (CTF) Through 36 Months
Description: Evaluated by assessing the rate of subjects free of chronic treatment failure with paroxysmal atrial fibrillation who have failed one or more Atrial Fibrillation Drugs (AFDs).
  Chronic treatment failure is defined as:
  * Documented atrial fibrillation lasting longer than 30 seconds (outside the 90 day blanking period) OR
  * Intervention for atrial fibrillation (except for repeat cryoablation during the 90 day blanking period)
Time Frame: Through 36 months
Population: Enrolled subjects that met all inclusion and no exclusion criteria, and who underwent a study cryoablation procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Modified Intent to Treat Group (mITT)
Number analyzed (Participants) | 354
Percentage of participants | 66.9 [61.6 to 71.7]
Statistical Analysis 1: Comparison: Modified Intent to Treat Group (mITT); Test type: Superiority; p < 0.001, Exact binomial; Exact binomial p-value is shown, but the confidence intervals reported are calculated from Greenwood's approximation of the standard error; Kaplan-Meier (product-limit) estimator = 66.9, 95% CI 2-sided [61.6 to 71.7]

2. Primary Outcome: Safety: Percentage of Participants Experiencing Cryoablation Procedure Events (CPEs) Through 12 Months
Description: Demonstrate safety (through 12 months) of Arctic Front® Cardiac CryoAblation Catheter System, including the Freezor® MAX Cardiac Cryoablation Catheter by assessing the rate of subjects experiencing Cryoablation Procedure Events (CPEs) with paroxysmal atrial fibrillation who have failed one or more Atrial Fibrillation Drugs (AFDs).
Time Frame: 12 Months
Population: Enrolled subjects that met all inclusion and no exclusion criteria, and who underwent a study cryoablation procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Modified Intent to Treat Group (mITT)
Number analyzed (Participants) | 354
Percentage of participants | 2.3 [1.1 to 4.5]
Statistical Analysis 1: Comparison: Modified Intent to Treat Group (mITT); Test type: Superiority; p < 0.001, Exact binomial; [statistical method as in outcome 1, analysis 1]; Kaplan-Meier (product-limit) estimator = 2.3, 95% CI 2-sided [1.1 to 4.5]

3. Secondary Outcome: Chronic Safety: Percentage of Participants Free From Major Atrial Fibrillation Events (MAFE) at 1, 2 and 3 Years.
Description: Freedom from Major Atrial Fibrillation Event (MAFE): A MAFE is a serious adverse event (SAE) which has not been categorized as a cryoablation procedure event.
Time Frame: Annually, through 3 years
Population: Enrolled subjects that met all inclusion and no exclusion criteria, and who underwent a study cryoablation procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Modified Intent to Treat Group (mITT)
Number analyzed (Participants) | 354
Percentage of participants
  Freedom from MAFEs in mITT subjects at 1 year | 90.3 [86.6 to 92.9]
  Freedom from MAFEs in mITT subjects at 2 years | 83.2 [78.8 to 86.8]
  Freedom from MAFEs in mITT subjects at 3 years | 77.8 [72.9 to 81.9]
Statistical Analysis 1: Comparison: Modified Intent to Treat Group (mITT); Test type: Other — Secondary analyses were exploratory. No formal hypotheses or performance criteria were predefined; Freedom from MAFE's was estimated using Kaplan-Meier methods

4. Secondary Outcome: Chronic Effectiveness: Percentage of Participants Free of Chronic Treatment Failure (CTF) at 1 and 2 Years
Description: Freedom from chronic treatment failure, defined as:
  * Documented atrial fibrillation lasting longer than 30 seconds (outside the 90 day blanking period) OR
  * Intervention for atrial fibrillation (except for repeat cryoablation during the 90 day blanking period)
Time Frame: Annually, at 1 and 2 years
Population: Enrolled subjects that met all inclusion and no exclusion criteria, and who underwent a study cryoablation procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Modified Intent to Treat Group (mITT)
Number analyzed (Participants) | 354
Percentage of participants
  1 year freedom from CTF | 80.4 [75.9 to 84.2]
  2 year freedom from CTF | 72.8 [67.7 to 77.2]
Statistical Analysis 1: Comparison: Modified Intent to Treat Group (mITT); Test type: Other — Secondary analyses were exploratory. No formal hypotheses or performance criteria were predefined; Chronic treatment success was estimated at one and two years using Kaplan-Meier methods

ADVERSE EVENTS:
Time Frame: All adverse events were collected between subject consent (enrollment) and study completion (3 years post study cryoablation procedure) or study exit.
Groups:
- Treated Group: Enrolled subjects who underwent a study cryoablation procedure whether or not they met all inclusion/exclusion criteria.
Arm/Group | Treated Group
All-Cause Mortality (participants affected / at risk) | 5/359
Serious Adverse Events (participants affected / at risk) | 145/359
Other Adverse Events (participants affected / at risk) | 70/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Group (N=359)
Atrial Fibrillation (Cardiac disorders) | 65 (75)
Atrial Flutter (Cardiac disorders) | 20 (20)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (9)
Coronary Artery Disease (Cardiac disorders) | 3 (5)
Urinary Tract Infection (Infections and infestations) | 5 (5)
Cardiac Failure Congestive (Cardiac disorders) | 4 (4)
Meniscus Injury (Injury, poisoning and procedural complications) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 3 (3)
Phrenic Nerve Paralysis (Nervous system disorders) | 3 (3)
Post procedural haemmorhage (Injury, poisoning and procedural complications) | 3 (3)
Sinus node dysfunction (Cardiac disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Angina Pectoris (Cardiac disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Chest pain (General disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haematoma (Vascular disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Accidental death (General disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
CHA2DS2-VASc annual stroke risk moderate (Investigations) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cerebral Haemmorhage (Nervous system disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colostomy closure (Surgical and medical procedures) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal haemmorhage (Gastrointestinal disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemmorhage intracranial (Nervous system disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Mitral valve calcification (Cardiac disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Nodal rhythym (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Post procedural bile leak (Hepatobiliary disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal haemmorhage (Gastrointestinal disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Group (N=359)
Atrial fibrillation (Cardiac disorders) | 70 (98)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (4):
  • Study Protocol: Clinical Investigation Plan Version 4 (2011-08-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT01456949/Prot_001.pdf
  • Study Protocol: Clinical Investigation Plan Version 5 (2013-09-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT01456949/Prot_002.pdf
  • Study Protocol: Clinical Investigation Plan Version 6 (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT01456949/Prot_003.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT01456949/SAP_000.pdf